CLINICAL TRIAL: NCT06058507
Title: "The Incidence of Carotid Web and Its Radiological Classification, Determination of Its Relationship With Ischemic Stroke by Evaluating the Clinical Data and Vascular Risk Factors of Carotid Web Cases"
Brief Title: "Carotid Web Incidence and Radiological Classification, Determination of Its Relationship With Ischemic Stroke"
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ekin Öykü Baylam Yirmibeş, RESEARCH ASSISTANT, Suleyman Demirel University
Other Study IDs: SDUWEB
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Stroke; Transient Ischemic Attack; Carotid Artery Diseases
Keywords: carotid web; ischemic stroke; transient ischemic atack
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Carotid Artery Diseases; Ischemic Stroke | interventions — Computed Tomography Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with carotid web detected: Patients in whom carotid web was detected by examining carotid CTA images
  Interventions: Diagnostic Test: CT angiography

INTERVENTIONS:
Diagnostic Test: CT angiography — No intervention was made

SUMMARY:
In our research, we aim to increase awareness on this issue by classifying the frequency of carotid webs and their radiological classification; Evaluating the clinical data and vascular risk factors of carotid web cases and determining their relationship with ischemic stroke and determining the measures that can be taken for future optimal treatment.

We aimed to contribute to their approach.

DETAILED DESCRIPTION:
Carotid web is a thin membrane-like tissue that extends from the wall to the lumen of the carotid artery bulb, identified radiologically. It is considered that stroke may be related to altered hemodynamics, blood stasis and fibrin-based clot embolization mechanisms in the distal carotid web. Radiologically, in DSA and CTA, there is a thin membrane-like intraluminal filling defect extending along the posterior carotid wall in oblique-sagittal sections and a corresponding defect in axial sections.

It is seen as a thin septum; There is no study on its classification in the literature. Determination of the incidence of carotid web, determination of its relationship with ischemic stroke / TİA, Facilitating distinctions such as dissection etc. by making radiological classification is important in terms of increasing awareness on this issue and early diagnosis. Demonstrating the relationship between carotid webs, which are shown as a cryptogenic cause of stroke, and vascular risk factors and taking protective measures against them will be effective in preventing strokes. In our research, we aim to increase awareness on this issue by classifying the frequency of carotid webs and their radiological classification; We aimed to evaluate the clinical data and vascular risk factors of carotid web cases, determine their relationship with ischemic stroke, and determine the precautions that can be taken to contribute to future optimal treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old

  * Having a preliminary diagnosis of cerebrovascular disease
  * Having carotid CTA and/or DSA imaging performed

Exclusion Criteria:

* Being under 18 years of age
* Patients who cannot undergo CTA and/or DSA imaging due to the risk of contrast material allergy or renal failure.
* Patients for whom consent for imaging cannot be obtained by the patient and their relatives and for whom CTA/DSA examination is not required in terms of etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who underwent carotid CTA and/or DSA imaging with the preliminary diagnosis of cerebrovascular disease and a carotid web was detected.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
ischemic stroke | 1 year
  dysarthria, weakness, facial paralysis

SECONDARY OUTCOMES:
transient ischemic atack | 1 year
  temporary weakness and slurred speech

CONTACTS AND LOCATIONS:
Overall Officials: ekin EB baylam yirmibeş, Principal Investigator — Suleyman Demirel University
Locations (1):
- Suleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No